CLINICAL TRIAL: NCT00191282
Title: Hyperglycemia and Its Effect After Acute Myocardial Infarction on Cardiovascular Outcomes in Patients With Type 2 Diabetes (HEART2D)
Brief Title: Hyperglycemia and Cardiovascular Outcomes With Type 2 Diabetes
Acronym: IONM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5509; F3Z-MC-IONM (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus, Type 2; Acute Myocardial Infarction
Keywords: diabetes; MI; heart attack
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Myocardial Infarction | interventions — Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Postprandial: Premeal insulin lispro +/- bedtime NPH
  Interventions: Drug: Insulin lispro; Drug: Human insulin isophane suspension (NPH)
- 2 (Active Comparator): Fasting: NPH/insulin glargine or human insulin 30/70
  Interventions: Drug: Insulin glargine; Drug: Human insulin isophane suspension; Drug: Human insulin 30/70

INTERVENTIONS:
Drug: Insulin lispro — Patient adjusted dose, three times a day (TID), injected subcutaneous (SC) before each meal until patient completes study
  Other Names: Humalog
  Arms: 1
Drug: Human insulin isophane suspension (NPH) — Patient adjusted dose, daily at bedtime, injected subcutaneous (SC) until patient completes study. To be added to the arm only if patient has two consecutive HbA1c values >8.0%
  Arms: 1
Drug: Insulin glargine — Insulin glargine injected subcutaneous (SC) once daily in the evening until patient completes study.
  Arms: 2
Drug: Human insulin isophane suspension — Patient adjusted dose, twice daily, injected subcutaneous (SC) before morning and evening meals until patient completes study.
  Arms: 2
Drug: Human insulin 30/70 — Patient adjusted dose, twice daily before the morning and evening meals, injected subcutaneous (SC) until patient completes study. To replace insulin regimen in this arm only if patient has two consecutive HbA1c values >8.0%.
  Other Names: Human insulin 70/30 (in the United States)
  Arms: 2

SUMMARY:
The primary objective was to demonstrate a difference between two insulin strategies, one targeting postprandial (PP) hyperglycemia and the other targeting fasting and interprandial hyperglycemia, on time until the first combined adjudicated cardiovascular (CV) event (primary outcome defined as CV death, nonfatal myocardial infarction [MI], nonfatal stroke, coronary revascularization, or hospitalized acute coronary syndrome).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of two different treatment strategies on CV outcomes in patients with type 2 diabetes while aiming to achieve and maintain HbA1c <7.0% in both groups. Only patients who have recently experienced an acute MI will be considered for participation in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 30 years old
* Have had type 2 diabetes for at least 3 months prior to Visit 1
* Were admitted to the Coronary Care Unit (CCU) within 18 days prior to Visit 1 for an acute MI
* Are capable and willing to do specified study procedures
* Have given informed consent to participate in the study in accordance with local regulations

Exclusion Criteria:

* Were on one of the following therapies prior to admission to the CCU for the recent MI: a)diet therapy only and have glycosylated hemoglobin (HbA1c) <1.15 times the upper limit of normal or b) an intensive basal/bolus insulin regimen
* Are using any oral antihyperglycemic medication at the time of Visit 2 and are unwilling to stop the use of such medication for the duration of the study
* Have substantial myocardial damage, which would significantly outweigh the potential benefit of the treatment strategies for diabetes
* Have the most severe form of congestive heart failure
* Have liver disease so severe that it precludes the patient from following and completing the protocol

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1116 (Actual)
Dates: Start 2002-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9am-5pm Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-651-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Toronto, Ontario, Canada
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-651-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Zagreb, Croatia
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-651-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Prague, Czechia
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-651-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Dresden, Germany
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-651-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Budapest, Hungary
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-651-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, New Delhi, India
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-651-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Jerusalem, Israel
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-651-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Beirut, Lebanon
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-651-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Warsaw, Poland
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-651-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Brasov, Romania
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-651-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Saint Petersburg, Russia
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-651-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Nitra, Slovakia
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-651-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Maribor, Slovenia
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-651-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Parktown, South Africa
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-651-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Barcelona, Spain
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-651-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Istanbul, Turkey (Türkiye)
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-651-4559), Monday-Friday, 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Liverpool, United Kingdom

REFERENCES:
- [Result] Raz I, Wilson PW, Strojek K, Kowalska I, Bozikov V, Gitt AK, Jermendy G, Campaigne BN, Kerr L, Milicevic Z, Jacober SJ. Effects of prandial versus fasting glycemia on cardiovascular outcomes in type 2 diabetes: the HEART2D trial. Diabetes Care. 2009 Mar;32(3):381-6. doi: 10.2337/dc08-1671. PMID 19246588
- [Result] Milicevic Z, Raz I, Beattie SD, Campaigne BN, Sarwat S, Gromniak E, Kowalska I, Galic E, Tan M, Hanefeld M. Natural history of cardiovascular disease in patients with diabetes: role of hyperglycemia. Diabetes Care. 2008 Feb;31 Suppl 2:S155-60. doi: 10.2337/dc08-s240. PMID 18227478
- [Result] Milicevic Z, Raz I, Strojek K, Skrha J, Tan MH, Wyatt JW, Beattie SD, Robbins DC; HEART2D Study. Hyperglycemia and its effect after acute myocardial infarction on cardiovascular outcomes in patients with Type 2 diabetes mellitus (HEART2D) Study design. J Diabetes Complications. 2005 Mar-Apr;19(2):80-7. doi: 10.1016/j.jdiacomp.2004.06.003. PMID 15745837
- [Derived] Raz I, Ceriello A, Wilson PW, Battioui C, Su EW, Kerr L, Jones CA, Milicevic Z, Jacober SJ. Post hoc subgroup analysis of the HEART2D trial demonstrates lower cardiovascular risk in older patients targeting postprandial versus fasting/premeal glycemia. Diabetes Care. 2011 Jul;34(7):1511-3. doi: 10.2337/dc10-2375. Epub 2011 May 18. PMID 21593301
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient was randomized but discontinued prior to treatment and is not included in any of the analyses. In the Participant Flow table, the term study outcome is used to differentiate it from serious adverse events (SAEs). By definition, the study outcomes were all SAEs as it was a cardiovascular outcome trial.
Groups:
- Postprandial: Insulin lispro: Patient adjusted dose, three times a day (TID), injected subcutaneous (SC) before each meal until patient completes study; Human insulin isophane suspension: Patient adjusted dose, daily at bedtime, injected subcutaneous (SC) until patient completes study. To be added to the arm only if patient has two consecutive HbA1c values >8.0%.
- Fasting: Human insulin isophane suspension: injected subcutaneous (SC) twice daily before the morning and evening meals until patient completes study; Insulin glargine: injected subcutaneous (SC) once daily in the evening until patient completes study; or Human insulin 30/70: Patient adjusted dose, twice daily before the morning and evening meals, injected subcutaneous (SC) until patient completes study. To replace insulin regimen in this arm only if patient has two consecutive HbA1c values >8.0%.
Period: Overall Study
Arm/Group | Postprandial | Fasting
Started | 558 | 558
Completed | 338 | 346
Not Completed | 220 | 212
Not completed — Adverse Event | 5 | 6
Not completed — Death | 51 | 51
Not completed — Lack of Efficacy | 11 | 6
Not completed — Noncompliance | 14 | 17
Not completed — Patient moved | 11 | 14
Not completed — Withdrawal by Subject | 59 | 44
Not completed — Physician Decision | 18 | 15
Not completed — Protocol entry criteria not met | 14 | 9
Not completed — Protocol Violation | 9 | 12
Not completed — Severity of outcome | 2 | 5
Not completed — Sponsor's decision | 2 | 2
Not completed — Lost to Follow-up | 24 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Postprandial | Fasting | Total
Number analyzed (Participants) | 557 | 558 | 1115
Age Continuous [Mean (Standard Deviation); unit: years] | 61.1 (9.7) | 60.9 (9.8) | 61.0 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 208 | 409
  Male | 356 | 350 | 706
Region of Enrollment [Number; unit: participants]
  Slovakia (Slovak Republic) | 8 | 11 | 19
  Slovenia | 16 | 16 | 32
  Spain | 5 | 3 | 8
  Lebanon | 18 | 19 | 37
  Turkey | 19 | 17 | 36
  Israel | 38 | 38 | 76
  Russian Federation | 63 | 65 | 128
  United Kingdom | 15 | 18 | 33
  India | 36 | 34 | 70
  Czech Republic | 26 | 24 | 50
  Hungary | 41 | 41 | 82
  Canada | 12 | 13 | 25
  Poland | 102 | 103 | 205
  Croatia | 72 | 71 | 143
  Romania | 33 | 31 | 64
  South Africa | 44 | 45 | 89
  Germany | 9 | 9 | 18
Race/Ethnicity [Number; unit: participants]
  Caucasian | 484 | 483 | 967
  Western Asian | 61 | 58 | 119
  African Descent | 1 | 6 | 7
  Other | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Primary Combined Outcome
Description: The combined study outcomes consisted of cardiovascular (CV) death, nonfatal myocardial infarction (MI), nonfatal stroke, hospitalization for acute coronary syndromes (HACS), and coronary revascularization procedures planned after randomization.
Time Frame: Randomization (Day 0) until first occurrence of primary combined outcome (18 month initial treatment period, extended treatment follow-up period up to 5.5 years)
Population: All randomized patients who took at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 557 | 558
participants | 174 | 181
Statistical Analysis 1: Comparison: Postprandial vs Fasting; To achieve 80% power, 490 pts need to experience primary combined CV outcome to detect diff. between treatments, assuming: >=18.5% reduction in incidence of outcomes, 18 mo. pt recruitment, 18 mo. pt follow-up, 10% annual drop-out rate, 2-yr outcome incidence rate of >=40% (pts in least efficacious treatment), and nominal 2-sided signif. of 0.045; Test type: Superiority or Other; p = 0.866, Log Rank; Hazard Ratio (HR) = 0.98

2. Secondary Outcome: Number of Participants Who Experienced Death From Any Cause or Any One of the Primary Outcomes
Description: Primary outcomes in this study consisted of: cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, hospitalization for acute coronary syndromes (HACS), and coronary revascularization procedure planned after randomization.
Time Frame: Randomization (Day 0) until death from any cause or one of the primary outcomes (18 month initial treatment period, extended treatment follow-up period up to 5.5 years)
Population: All randomized patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 557 | 558
participants | 178 | 189
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.715, Log Rank; Hazard Ratio (HR) = 0.96

3. Secondary Outcome: Number of Participants Who Experienced Any One of the Primary Outcomes Adjusted for Indicators of Metabolic Control
Description: Indicators of metabolic control included glycosylated hemoglobin (HbA1c) and fasting blood glucose concentrations.
Time Frame: Randomization (Day 0) until occurrence of primary outcome (18 month initial treatment period, extended treatment follow-up period up to 5.5 years)
Population: All randomized patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 557 | 558
participants | 174 | 181
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.914, Log Rank; Hazard Ratio (HR) = 1.01

4. Secondary Outcome: Number of Participants Who Experienced Primary Outcomes Adjusted for Metabolic Control and Major Cardiovascular (CV) Risk Factors
Description: Primary outcomes adjusted for major cardiovascular (CV) risk factors (blood pressure, cholesterol [total, high density lipoprotein (HDL), and low density lipoprotein (LDL)], triglycerides, smoking, albuminuria, age, gender, and body mass index (BMI).
Time Frame: as for outcome 3
Population: All randomized patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 557 | 558
participants | 174 | 181
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.706, Log Rank; Hazard Ratio (HR) = 1.05

5. Secondary Outcome: Number of Participants Who Experienced Death From Any Cause
Time Frame: Randomization (Day 0) until death from any cause (18 month initial treatment period, extended treatment follow-up period up to 5.5 years)
Population: All randomized patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 557 | 558
participants | 51 | 51
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.982, Log Rank; Hazard Ratio (HR) = 1.00

6. Secondary Outcome: Number of Participants Who Experienced Cardiovascular (CV) Death
Time Frame: Randomization (Day 0) until cardiovascular death (18 month initial treatment period, extended treatment follow-up period up to 5.5 years)
Population: All randomized patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 557 | 558
participants | 44 | 42
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.816, Log Rank; Hazard Ratio (HR) = 1.05

7. Secondary Outcome: Number of Participants Who Experienced Myocardial Infarction (MI)
Description: Occurrence of myocardial infarction (MI) (fatal, nonfatal, any).
Time Frame: Randomization (Day 0) until myocardial infarction (18 month initial treatment period, extended treatment follow-up period up to 5.5 years)
Population: All randomized patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 557 | 558
participants | 63 | 63
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.948, Log Rank; Hazard Ratio (HR) = 1.01

8. Secondary Outcome: Number of Participants Who Experienced Stroke
Description: Occurrence of stroke (fatal, nonfatal, any).
Time Frame: Randomization (Day 0) until stroke (18 month initial treatment period, extended treatment follow-up period up to 5.5 years)
Population: All randomized patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 557 | 558
participants | 20 | 17
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.581, Log Rank; Hazard Ratio (HR) = 1.20

9. Secondary Outcome: Number of Participants Who Experienced Hospitalization for Acute Coronary Syndromes (HACS)
Time Frame: Randomization (Day 0) until HACS (18 month initial treatment period, extended treatment follow-up period up to 5.5 years)
Population: All randomized patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 557 | 558
participants | 58 | 54
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.647, Log Rank; Hazard Ratio (HR) = 1.09

10. Secondary Outcome: Number of Participants Who Experienced Coronary Revascularization Procedures
Description: Occurrence of all coronary revascularization procedures (angioplasty or coronary artery by-pass surgery) planned after randomization.
Time Frame: Randomization (Day 0) until coronary revascularization procedures (18 month initial treatment period, extended treatment follow-up period up to 5.5 years)
Population: All randomized patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 557 | 558
participants | 84 | 94
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.525, Log Rank; Hazard Ratio (HR) = 0.91

11. Secondary Outcome: Number of Participants Who Experienced Amputation for Peripheral Vascular Disease Planned After Randomization
Time Frame: Randomization (Day 0) until amputation (18 month initial treatment period, extended treatment follow-up period up to 5.5 years)
Population: All randomized patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 557 | 558
participants | 9 | 8
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.800, Log Rank; Hazard Ratio (HR) = 1.13

12. Secondary Outcome: Number of Participants Who Experienced Congestive Heart Failure
Description: Occurrence of congestive heart failure (newly diagnosed after Visit 2).
Time Frame: Randomization (Day 0) until congestive heart failure (18 month initial treatment period, extended treatment follow-up period up to 5.5 years)
Population: All randomized patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 557 | 558
participants | 33 | 37
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.662, Log Rank; Hazard Ratio (HR) = 0.90

13. Secondary Outcome: Number of Participants Who Experienced Revascularization Procedure for Peripheral Vascular Disease Planned After Randomization
Time Frame: Randomization (Day 0) until revascularization procedure (18 month initial treatment period, extended treatment follow-up period up to 5.5 years)
Population: All randomized patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 557 | 558
participants | 11 | 12
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.863, Log Rank; Hazard Ratio (HR) = 0.93

14. Secondary Outcome: Number of Participants Who Experienced Coronary Angiography Planned After Randomization
Time Frame: Randomization (Day 0) until coronary angiography (18 month initial treatment period, extended treatment follow-up period up to 5.5 years)
Population: All randomized patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 557 | 558
participants | 75 | 86
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.471, Log Rank; Hazard Ratio (HR) = 0.89

15. Secondary Outcome: Number of Participants With Self-Reported Hypoglycemia During Month 1
Description: Hypoglycemia was defined as any time a patient feels, or another person observes, that the patient is experiencing a sign/symptom which he/she would associate with hypoglycemia (for example, tremors, headache, sweating, disorientation, weakness, etc) or a blood glucose measurement less than 3.5 mmol/L (63 mg/dL).
Time Frame: Visit 3 (Month 1)
Population: All randomized patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 557 | 557
participants | 124 | 119
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.7168, Chi-squared

16. Secondary Outcome: Number of Episodes of Self-Reported Hypoglycemia Reported by Participants With Self-Reported Hypoglycemia During Month 1
Description: as for outcome 15
Time Frame: Visit 3 (Month 1)
Population: All randomized participants who self-reported hypoglycemia during Month 1.
Measure: Number; unit: episodes of hypoglycemia
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 124 | 119
episodes of hypoglycemia | 353 | 302

17. Secondary Outcome: Number of Participants With Self-Reported Hypoglycemia During Month 3
Description: as for outcome 15
Time Frame: Visit 4 (Month 3)
Population: All randomized patients who took at least one dose of study drug and who were still in the study.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 511 | 525
participants | 160 | 139
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.0860, Chi-squared

18. Secondary Outcome: Number of Episodes of Self-Reported Hypoglycemia Reported by Participants With Self-Reported Hypoglycemia During Month 3
Description: as for outcome 15
Time Frame: Visit 4 (Month 3)
Population: All randomized participants who self-reported hypoglycemia during Month 3.
Measure: Number; unit: episodes of hypoglycemia
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 160 | 139
episodes of hypoglycemia | 567 | 524

19. Secondary Outcome: Number of Participants With Self-Reported Hypoglycemia During Month 6
Description: as for outcome 15
Time Frame: Visit 5 (Month 6)
Population: All randomized patients who took at least one dose of study drug and who were still in the study.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 493 | 504
participants | 163 | 145
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.1424, Chi-squared

20. Other Pre Specified Outcome: Summary of Reasons for Deaths
Time Frame: Randomization (Day 0) to death (18 month initial treatment period, extended treatment follow-up period up to 5.5 years)
Population: All randomized patients who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 557 | 558
participants
  Fatal MI | 12 | 12
  Fatal Stroke | 3 | 2
  CV Death other than Stroke/MI | 29 | 28
  Non-CV Death | 7 | 8
  Unknown | 0 | 1

21. Secondary Outcome: Number of Episodes of Self-Reported Hypoglycemia Reported by Participants With Self-Reported Hypoglycemia During Month 6
Description: as for outcome 15
Time Frame: Visit 5 (Month 6)
Population: All randomized participants with self-reported hypoglycemia during Month 6.
Measure: Number; unit: episodes of hypoglycemia
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 163 | 145
episodes of hypoglycemia | 770 | 576

22. Secondary Outcome: Number of Participants With Self-Reported Hypoglycemia During Month 9
Description: as for outcome 15
Time Frame: Visit 6 (Month 9)
Population: All randomized patients who took at least one dose of study drug and who were still in the study.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 483 | 488
participants | 155 | 138
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.1957, Chi-squared

23. Secondary Outcome: Number of Episodes of Self-Reported Hypoglycemia Reported by Participants With Self-Reported Hypoglycemia During Month 9
Description: as for outcome 15
Time Frame: Visit 6 (Month 9)
Population: All randomized participants with self-reported hypoglycemia during Month 9.
Measure: Number; unit: episodes of hypoglycemia
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 155 | 138
episodes of hypoglycemia
  Number of Episodes | 747 | 569

24. Secondary Outcome: Number of Participants With Self-Reported Hypoglycemia During Month 12
Description: as for outcome 15
Time Frame: Visit 7 (Month 12)
Population: All randomized patients who took at least one dose of study drug and who were still in the study.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 470 | 471
participants | 146 | 130
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.2434, Chi-squared

25. Secondary Outcome: Number of Episodes of Self-Reported Hypoglycemia Reported by Participants With Self-Reported Hypoglycemia During Month 12
Description: as for outcome 15
Time Frame: Visit 7 (Month 12)
Population: All randomized participants with self-reported hypoglycemia during Month 12.
Measure: Number; unit: episodes of hypoglycemia
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 146 | 130
episodes of hypoglycemia | 710 | 486

26. Secondary Outcome: Number of Participants With Self-Reported Hypoglycemia During Month 18
Description: as for outcome 15
Time Frame: Visit 8 (Month 18)
Population: All randomized patients who took at least one dose of study drug and who were still in the study.
Measure: Number; unit: participants
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 452 | 457
participants | 143 | 129
Statistical Analysis 1: Comparison: Postprandial vs Fasting; Test type: Superiority or Other; p = 0.2617, Chi-squared

27. Secondary Outcome: Number of Episodes of Self-Reported Hypoglycemia Reported by Participants With Self-Reported Hypoglycemia During Month 18
Description: as for outcome 15
Time Frame: Visit 8 (Month 18)
Population: All randomized participants with self-reported hypoglycemia during Month 18.
Measure: Number; unit: episodes of hypoglycemia
Arm/Group | Postprandial | Fasting
Number analyzed (Participants) | 143 | 129
episodes of hypoglycemia | 945 | 669

ADVERSE EVENTS:
Arm/Group | Postprandial | Fasting
Serious Adverse Events (participants affected / at risk) | 145 | 142
Other Adverse Events (participants affected / at risk) | 356 | 346
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Postprandial | Fasting
Anaemia (Blood and lymphatic system disorders) | 1/557 (1) | 1/558 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1/557 (1) | 0/558 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0/557 (0) | 1/558 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1/557 (1) | 0/558 (0)
Acute coronary syndrome (Cardiac disorders) | 0/557 (0) | 1/558 (1)
Acute left ventricular failure (Cardiac disorders) | 1/557 (1) | 0/558 (0)
Acute myocardial infarction (Cardiac disorders) | 0/557 (0) | 2/558 (2)
Angina pectoris (Cardiac disorders) | 3/557 (3) | 3/558 (3)
Angina unstable (Cardiac disorders) | 2/557 (2) | 1/558 (1)
Atrial fibrillation (Cardiac disorders) | 2/557 (2) | 7/558 (7)
Atrial flutter (Cardiac disorders) | 1/557 (1) | 0/558 (0)
Atrioventricular block (Cardiac disorders) | 0/557 (0) | 1/558 (1)
Atrioventricular block complete (Cardiac disorders) | 0/557 (0) | 1/558 (1)
Atrioventricular block second degree (Cardiac disorders) | 1/557 (1) | 0/558 (0)
Cardiac failure (Cardiac disorders) | 2/557 (2) | 1/558 (1)
Cardiac failure chronic (Cardiac disorders) | 0/557 (0) | 2/558 (2)
Cardiac failure congestive (Cardiac disorders) | 8/557 (8) | 8/558 (8)
Conduction disorder (Cardiac disorders) | 1/557 (1) | 0/558 (0)
Coronary artery insufficiency (Cardiac disorders) | 0/557 (0) | 1/558 (1)
Coronary artery restenosis (Cardiac disorders) | 1/557 (1) | 0/558 (0)
Dressler's syndrome (Cardiac disorders) | 0/557 (0) | 1/558 (1)
Intracardiac thrombus (Cardiac disorders) | 0/557 (0) | 1/558 (1)
Left ventricular dysfunction (Cardiac disorders) | 0/557 (0) | 1/558 (1)
Left ventricular failure (Cardiac disorders) | 0/557 (0) | 1/558 (1)
Mitral valve incompetence (Cardiac disorders) | 1/557 (1) | 0/558 (0)
Myocardial infarction (Cardiac disorders) | 1/557 (1) | 2/558 (2)
Sick sinus syndrome (Cardiac disorders) | 2/557 (2) | 2/558 (2)
Sinus bradycardia (Cardiac disorders) | 1/557 (1) | 0/558 (0)
Ventricular extrasystoles (Cardiac disorders) | 0/557 (0) | 1/558 (1)
Ventricular fibrillation (Cardiac disorders) | 1/557 (1) | 0/558 (0)
Ventricular tachyarrhythmia (Cardiac disorders) | 0/557 (0) | 1/558 (1)
Ventricular tachycardia (Cardiac disorders) | 2/557 (2) | 1/558 (1)
Hearing impaired (Ear and labyrinth disorders) | 0/557 (0) | 1/558 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 0/557 (0) | 1/558 (1)
Vertigo (Ear and labyrinth disorders) | 2/557 (2) | 0/558 (0)
Vestibular neuronitis (Ear and labyrinth disorders) | 1/557 (1) | 0/558 (0)
Hyperthyroidism (Endocrine disorders) | 1/557 (1) | 0/558 (0)
Cataract (Eye disorders) | 3/557 (3) | 1/558 (1)
Conjunctivitis (Eye disorders) | 0/557 (0) | 1/558 (1)
Diabetic retinopathy (Eye disorders) | 2/557 (2) | 1/558 (1)
Glaucoma (Eye disorders) | 0/557 (0) | 1/558 (1)
Retinal detachment (Eye disorders) | 1/557 (1) | 0/558 (0)
Vitreous haemorrhage (Eye disorders) | 1/557 (1) | 0/558 (0)
Abdominal pain (Gastrointestinal disorders) | 2/557 (2) | 2/558 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1/557 (1) | 2/558 (2)
Anal haemorrhage (Gastrointestinal disorders) | 1/557 (1) | 0/558 (0)
Colonic polyp (Gastrointestinal disorders) | 1/557 (1) | 1/558 (1)
Diarrhoea (Gastrointestinal disorders) | 1/557 (1) | 1/558 (1)
Duodenitis (Gastrointestinal disorders) | 1/557 (1) | 0/558 (0)
Dyspepsia (Gastrointestinal disorders) | 0/557 (0) | 1/558 (1)
Enteritis (Gastrointestinal disorders) | 1/557 (1) | 0/558 (0)
Enterocolitis (Gastrointestinal disorders) | 0/557 (0) | 1/558 (1)
Gastric polyps (Gastrointestinal disorders) | 0/557 (0) | 1/558 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1/557 (1) | 0/558 (0)
Gastritis (Gastrointestinal disorders) | 3/557 (3) | 2/558 (2)
Gastritis erosive (Gastrointestinal disorders) | 0/557 (0) | 1/558 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2/557 (2) | 0/558 (0)
Gastrointestinal telangiectasia (Gastrointestinal disorders) | 1/557 (1) | 0/558 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0/557 (0) | 2/558 (2)
Haemorrhoids (Gastrointestinal disorders) | 1/557 (1) | 1/558 (1)
Hiatus hernia (Gastrointestinal disorders) | 1/557 (1) | 2/558 (2)
Ileus (Gastrointestinal disorders) | 1/557 (1) | 0/558 (0)
Inguinal hernia (Gastrointestinal disorders) | 2/557 (2) | 0/558 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0/557 (0) | 1/558 (1)
Melaena (Gastrointestinal disorders) | 0/557 (0) | 2/558 (2)
Mouth cyst (Gastrointestinal disorders) | 0/557 (0) | 1/558 (1)
Nausea (Gastrointestinal disorders) | 1/557 (1) | 1/558 (1)
Peptic ulcer (Gastrointestinal disorders) | 1/557 (1) | 0/558 (0)
Peritonitis (Gastrointestinal disorders) | 1/557 (1) | 0/558 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0/557 (0) | 1/558 (1)
Vomiting (Gastrointestinal disorders) | 0/557 (0) | 2/558 (2)
Asthenia (General disorders) | 2/557 (2) | 1/558 (1)
Chest discomfort (General disorders) | 1/557 (1) | 1/558 (1)
Chest pain (General disorders) | 4/557 (4) | 6/558 (6)
Cyst (General disorders) | 0/557 (0) | 1/558 (1)
Hernia obstructive (General disorders) | 0/557 (0) | 1/558 (1)
Multi-organ failure (General disorders) | 1/557 (1) | 2/558 (2)
Non-cardiac chest pain (General disorders) | 2/557 (2) | 2/558 (2)
Oedema peripheral (General disorders) | 1/557 (1) | 0/558 (0)
Pyrexia (General disorders) | 3/557 (3) | 1/558 (1)
Bile duct stone (Hepatobiliary disorders) | 0/557 (0) | 2/558 (2)
Biliary colic (Hepatobiliary disorders) | 0/557 (0) | 1/558 (1)
Cholangitis (Hepatobiliary disorders) | 0/557 (0) | 1/558 (1)
Cholecystitis (Hepatobiliary disorders) | 1/557 (1) | 1/558 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1/557 (1) | 1/558 (1)
Cholelithiasis (Hepatobiliary disorders) | 1/557 (1) | 3/558 (3)
Hepatic cirrhosis (Hepatobiliary disorders) | 1/557 (1) | 0/558 (0)
Hypersensitivity (Immune system disorders) | 1/557 (1) | 0/558 (0)
Sarcoidosis (Immune system disorders) | 0/557 (0) | 1/558 (1)
Abscess limb (Infections and infestations) | 0/557 (0) | 1/558 (1)
Abscess neck (Infections and infestations) | 0/557 (0) | 1/558 (1)
Appendicitis (Infections and infestations) | 2/557 (2) | 2/558 (2)
Arthritis bacterial (Infections and infestations) | 0/557 (0) | 1/558 (1)
Bronchitis (Infections and infestations) | 3/557 (3) | 3/558 (3)
Bronchopneumonia (Infections and infestations) | 0/557 (0) | 3/558 (3)
Campylobacter gastroenteritis (Infections and infestations) | 0/557 (0) | 1/558 (1)
Cellulitis (Infections and infestations) | 3/557 (3) | 3/558 (3)
Chronic tonsillitis (Infections and infestations) | 0/557 (0) | 1/558 (1)
Diverticulitis (Infections and infestations) | 0/557 (0) | 1/558 (1)
Erysipelas (Infections and infestations) | 1/557 (1) | 1/558 (1)
Gangrene (Infections and infestations) | 1/557 (1) | 0/558 (0)
Gastroenteritis (Infections and infestations) | 1/557 (1) | 2/558 (2)
Intervertebral discitis (Infections and infestations) | 1/557 (1) | 0/558 (0)
Localised infection (Infections and infestations) | 1/557 (1) | 0/558 (0)
Lower respiratory tract infection (Infections and infestations) | 1/557 (1) | 2/558 (2)
Mediastinitis (Infections and infestations) | 1/557 (1) | 0/558 (0)
Meningitis (Infections and infestations) | 1/557 (1) | 0/558 (0)
Meningitis aseptic (Infections and infestations) | 1/557 (1) | 0/558 (0)
Nasopharyngitis (Infections and infestations) | 1/557 (1) | 0/558 (0)
Osteomyelitis (Infections and infestations) | 1/557 (1) | 0/558 (0)
Paronychia (Infections and infestations) | 0/557 (0) | 1/558 (1)
Perianal abscess (Infections and infestations) | 0/557 (0) | 1/558 (1)
Pneumonia (Infections and infestations) | 7/557 (7) | 4/558 (4)
Postoperative wound infection (Infections and infestations) | 1/557 (1) | 1/558 (1)
Purulent pericarditis (Infections and infestations) | 0/557 (0) | 1/558 (1)
Pyelonephritis (Infections and infestations) | 0/557 (0) | 1/558 (1)
Pyelonephritis chronic (Infections and infestations) | 0/557 (0) | 1/558 (1)
Pyometra (Infections and infestations) | 0/557 (0) | 1/558 (1)
Respiratory tract infection viral (Infections and infestations) | 0/557 (0) | 1/558 (1)
Sepsis (Infections and infestations) | 5/557 (5) | 0/558 (0)
Septic arthritis staphylococcal (Infections and infestations) | 0/557 (0) | 1/558 (1)
Septic shock (Infections and infestations) | 2/557 (2) | 2/558 (2)
Streptococcal bacteraemia (Infections and infestations) | 1/557 (1) | 0/558 (0)
Subcutaneous abscess (Infections and infestations) | 0/557 (0) | 1/558 (1)
Urinary tract infection (Infections and infestations) | 5/557 (5) | 4/558 (4)
Wound infection (Infections and infestations) | 1/557 (1) | 0/558 (0)
Wound sepsis (Infections and infestations) | 3/557 (3) | 0/558 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1/557 (1) | 1/558 (1)
Excoriation (Injury, poisoning and procedural complications) | 1/557 (1) | 0/558 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2/557 (2) | 0/558 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1/557 (1) | 0/558 (0)
Glaucoma traumatic (Injury, poisoning and procedural complications) | 1/557 (1) | 0/558 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1/557 (1) | 0/558 (0)
Head injury (Injury, poisoning and procedural complications) | 0/557 (0) | 1/558 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0/557 (0) | 1/558 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1/557 (1) | 0/558 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1/557 (1) | 0/558 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0/557 (0) | 1/558 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0/557 (0) | 1/558 (1)
Blood pressure increased (Investigations) | 1/557 (1) | 0/558 (0)
Hepatic enzyme increased (Investigations) | 1/557 (1) | 0/558 (0)
International normalised ratio increased (Investigations) | 0/557 (0) | 1/558 (1)
Troponin increased (Investigations) | 1/557 (1) | 0/558 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1/557 (1) | 0/558 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4/557 (4) | 1/558 (1)
Diabetic foot (Metabolism and nutrition disorders) | 3/557 (3) | 1/558 (1)
Gout (Metabolism and nutrition disorders) | 1/557 (1) | 0/558 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4/557 (4) | 1/558 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1/557 (1) | 0/558 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 6/557 (6) | 7/558 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 0/557 (0) | 1/558 (1)
Insulin resistance (Metabolism and nutrition disorders) | 1/557 (1) | 0/558 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1/557 (1) | 0/558 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1/557 (1) | 0/558 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0/557 (0) | 1/558 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1/557 (1) | 1/558 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2/557 (2) | 0/558 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2/557 (2) | 0/558 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1/557 (1) | 0/558 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1/557 (1) | 0/558 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/557 (0) | 1/558 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/557 (0) | 1/558 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/557 (1) | 0/558 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/557 (1) | 0/558 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/557 (1) | 0/558 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/557 (1) | 0/558 (0)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/557 (1) | 0/558 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/557 (0) | 1/558 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/557 (1) | 1/558 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/557 (0) | 1/558 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/557 (1) | 0/558 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/557 (0) | 1/558 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/557 (2) | 0/558 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/557 (0) | 1/558 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/557 (0) | 1/558 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/557 (0) | 1/558 (1)
Renal cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/557 (0) | 1/558 (1)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/557 (1) | 0/558 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/557 (0) | 1/558 (1)
Amnesia (Nervous system disorders) | 0/557 (0) | 1/558 (1)
Carotid artery occlusion (Nervous system disorders) | 1/557 (1) | 0/558 (0)
Carotid artery stenosis (Nervous system disorders) | 2/557 (2) | 1/558 (1)
Cervicobrachial syndrome (Nervous system disorders) | 0/557 (0) | 1/558 (1)
Cluster headache (Nervous system disorders) | 0/557 (0) | 1/558 (1)
Diabetic neuropathy (Nervous system disorders) | 0/557 (0) | 1/558 (1)
Dizziness (Nervous system disorders) | 0/557 (0) | 1/558 (1)
Epilepsy (Nervous system disorders) | 0/557 (0) | 1/558 (1)
Headache (Nervous system disorders) | 1/557 (1) | 0/558 (0)
Hemiparesis (Nervous system disorders) | 0/557 (0) | 1/558 (1)
Hypotonia (Nervous system disorders) | 0/557 (0) | 1/558 (1)
Intercostal neuralgia (Nervous system disorders) | 1/557 (1) | 0/558 (0)
Mononeuropathy multiplex (Nervous system disorders) | 1/557 (1) | 0/558 (0)
Parkinson's disease (Nervous system disorders) | 1/557 (1) | 0/558 (0)
Presyncope (Nervous system disorders) | 1/557 (1) | 0/558 (0)
Psychomotor hyperactivity (Nervous system disorders) | 1/557 (1) | 0/558 (0)
Radiculopathy (Nervous system disorders) | 0/557 (0) | 1/558 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0/557 (0) | 1/558 (1)
Syncope (Nervous system disorders) | 2/557 (2) | 7/558 (7)
Transient ischaemic attack (Nervous system disorders) | 4/557 (4) | 0/558 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0/557 (0) | 1/558 (1)
Mood disorder due to a general medical condition (Psychiatric disorders) | 1/557 (1) | 0/558 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0/557 (0) | 1/558 (1)
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 1/557 (1) | 0/558 (0)
Calculus ureteric (Renal and urinary disorders) | 0/557 (0) | 1/558 (1)
Diabetic nephropathy (Renal and urinary disorders) | 1/557 (1) | 0/558 (0)
Haematuria (Renal and urinary disorders) | 0/557 (0) | 1/558 (1)
Renal artery stenosis (Renal and urinary disorders) | 1/557 (1) | 0/558 (0)
Renal colic (Renal and urinary disorders) | 0/557 (0) | 1/558 (1)
Renal failure (Renal and urinary disorders) | 2/557 (2) | 2/558 (2)
Renal failure acute (Renal and urinary disorders) | 1/557 (1) | 3/558 (3)
Renal failure chronic (Renal and urinary disorders) | 1/557 (1) | 2/558 (2)
Urethral obstruction (Renal and urinary disorders) | 0/557 (0) | 1/558 (1)
Urinary retention (Renal and urinary disorders) | 0/557 (0) | 1/558 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 2/557 (2) | 0/558 (0)
Polycystic ovaries (Reproductive system and breast disorders) | 0/557 (0) | 1/558 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0/557 (0) | 1/558 (1)
Uterine polyp (Reproductive system and breast disorders) | 1/557 (1) | 0/558 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1/557 (1) | 0/558 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1/557 (1) | 0/558 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/557 (1) | 0/558 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0/557 (0) | 1/558 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0/557 (0) | 3/558 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/557 (1) | 1/558 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1/557 (1) | 0/558 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0/557 (0) | 1/558 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1/557 (1) | 0/558 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0/557 (0) | 3/558 (3)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0/557 (0) | 1/558 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/557 (0) | 1/558 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3/557 (3) | 2/558 (2)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0/557 (0) | 1/558 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0/557 (0) | 1/558 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0/557 (0) | 1/558 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1/557 (1) | 0/558 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1/557 (1) | 0/558 (0)
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 0/557 (0) | 1/558 (1)
Photodermatosis (Skin and subcutaneous tissue disorders) | 0/557 (0) | 1/558 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1/557 (1) | 1/558 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 0/557 (0) | 1/558 (1)
Toe amputation (Surgical and medical procedures) | 1/557 (1) | 0/558 (0)
Accelerated hypertension (Vascular disorders) | 1/557 (1) | 0/558 (0)
Aortic aneurysm (Vascular disorders) | 1/557 (1) | 2/558 (2)
Arterial stenosis limb (Vascular disorders) | 0/557 (0) | 1/558 (1)
Arteriosclerosis obliterans (Vascular disorders) | 1/557 (1) | 0/558 (0)
Deep vein thrombosis (Vascular disorders) | 1/557 (1) | 0/558 (0)
Embolism (Vascular disorders) | 1/557 (1) | 0/558 (0)
Extremity necrosis (Vascular disorders) | 0/557 (0) | 1/558 (1)
Hypertension (Vascular disorders) | 2/557 (2) | 1/558 (1)
Hypertensive crisis (Vascular disorders) | 1/557 (1) | 0/558 (0)
Hypotension (Vascular disorders) | 1/557 (1) | 0/558 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 2/557 (2) | 1/558 (1)
Peripheral embolism (Vascular disorders) | 0/557 (0) | 1/558 (1)
Peripheral ischaemia (Vascular disorders) | 1/557 (1) | 0/558 (0)
Post thrombotic syndrome (Vascular disorders) | 1/557 (1) | 0/558 (0)
Shock (Vascular disorders) | 1/557 (1) | 0/558 (0)
Thrombosis (Vascular disorders) | 0/557 (0) | 1/558 (1)
Varicose vein (Vascular disorders) | 0/557 (0) | 1/558 (1)
Venous thrombosis (Vascular disorders) | 1/557 (1) | 0/558 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Postprandial | Fasting
Angina pectoris (Cardiac disorders) | 17/557 (17) | 22/558 (22)
Diabetic retinopathy (Eye disorders) | 25/557 (25) | 29/558 (29)
Chest pain (General disorders) | 19/557 (19) | 17/558 (17)
Oedema peripheral (General disorders) | 28/557 (28) | 28/558 (28)
Bronchitis (Infections and infestations) | 22/557 (22) | 23/558 (23)
Influenza (Infections and infestations) | 19/557 (19) | 29/558 (29)
Nasopharyngitis (Infections and infestations) | 35/557 (35) | 36/558 (36)
Urinary tract infection (Infections and infestations) | 14/557 (14) | 19/558 (19)
Arteriogram coronary (Investigations) | 25/557 (25) | 22/558 (22)
Weight increased (Investigations) | 19/557 (19) | 16/558 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20/557 (20) | 23/558 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 21/557 (21) | 28/558 (28)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9/557 (9) | 19/558 (19)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19/557 (19) | 25/558 (25)
Diabetic neuropathy (Nervous system disorders) | 23/557 (23) | 23/558 (23)
Headache (Nervous system disorders) | 19/557 (19) | 18/558 (18)
Depression (Psychiatric disorders) | 20/557 (20) | 13/558 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 27/557 (27) | 23/558 (23)
Hypertension (Vascular disorders) | 30/557 (30) | 27/558 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days